CLINICAL TRIAL: NCT06312800
Title: Acamprosate and Methazolamide for Essential Tremor: a Randomized Clinical Trial
Brief Title: Acamprosate and Methazolamide for Essential Tremor
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never initiated.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Peter LeWitt MD, Movement Disorder Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: LeWitt02
Record Dates: First submitted 2015-07-13; First posted 2024-03-15 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Essential Tremor
Keywords: Essential Tremor
MeSH Terms: conditions — Essential Tremor | interventions — Acamprosate; Methazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acamprosate (Experimental): Commercially available Acamprosate 333 mg tablets will be administered three times daily. Subjects will be started with one tablet with breakfast for 3 days, then one tablet with breakfast and dinner for 3 days, then one tablet 3 times a day for the next 15 days. Intervention order of medication trials will be determined by biostatistician.
  Interventions: Drug: Acamprosate
- Placebo (Active Comparator): Placebo tablets are not available from the manufacturer for either of these drugs which are marketed as white tablets about the size of an aspirin tablet. Custom made placebo tablets will be purchased that are about that size. While not ideal , the extent of disguising the drug identity should be adequate with this. The placebo tablets will be administered three times daily. Subjects will be started with one tablet with breakfast for 3 days, then one tablet with breakfast and dinner for 3 days, then one tablet 3 times a day for the next 15 days. Intervention order of medication trials will be determined by biostatistician
  Interventions: Drug: Placebo
- Methazolamide (Experimental): Commercially available methazolamide 50 mg tablets will be administered three times daily. Subjects will be started with one tablet with breakfast for 3 days, then one tablet with breakfast and dinner for 3 days, then one tablet 3 times a day for the next 15 days. Intervention order of medication trials will be determined by biostatistician
  Interventions: Drug: Methazolamide

INTERVENTIONS:
Drug: Acamprosate — Randomized allocation of treatments will guide the dispensation of treatments in one of 6 possible sequences--ex, M (methazolamide)- P(placebo)-A (Acamprosate); or PAM or MAP or PMA or AMP or APM. Biostatistician will devise medication randomization strategies and investigators and staff will be blinded.
  Arms: Acamprosate
Drug: Placebo — Randomized allocation of treatments will guide the dispensation of treatments in one of 6 possible sequences--ex, M (methazolamide)- P(placebo)-A (Acamprosate); or PAM or MAP or PMA or AMP or APM. Biostatistician will devise medication randomization strategies and investigators and staff will be blinded.
  Arms: Placebo
Drug: Methazolamide — Randomized allocation of treatments will guide the dispensation of treatments in one of 6 possible sequences--ex, M (methazolamide)- P(placebo)-A (Acamprosate); or PAM or MAP or PMA or AMP or APM. Biostatistician will devise medication randomization strategies and investigators and staff will be blinded.
  Arms: Methazolamide

SUMMARY:
This is an investigator initiated study is designed to evaluate the anti-tremor benefits of two marketed medications, methazolamide and acamprosate in subjects with a diagnosis of essential tremor (ET).

DETAILED DESCRIPTION:
This is an investigator-initiated study is designed to evaluate the anti-tremor benefits of two marketed medications, methazolamide and acamprosate in subjects with a diagnosis of essential tremor (ET). Methazolamide is approved by the FDA to treat glaucoma. Acamprosate is approved by the FDA and used in the treatment of alcoholism. Some subjects using these medications for those indications incidentally reported that they had improvement in their essential tremor symptoms.

The primary objective of this study is the change in the upper extremity tremor scores assessed by one of the tremor rating scales (FTMRS) compared to baseline. This scale has been used in previous reported studies. Secondary objectives will be to evaluate the change in the ratings on several scales between placebo and study medication treatment. Additionally, tremor amplitude will be measured with device called Kinesia HomeView. This has a sensor unit that is slipped over a finger and transmits information to a nearby computer. This device has been used by our staff in other clinical studies at our site to evaluate tremor symptoms.

The study is a double blind, parallel design with three separate treatment arms, each 3 weeks long . One arm is placebo, the other two are conventional dosing of either acamprosate (333 mg tablets TID) or methazolamide (50 mg tablets TID). Subjects who have ET and meet criteria will be randomized in varied order to undergo all three treatments. There will be a one-week washout period between arms of study treatments where subject are not on any study medication. Subjects who qualify will be titrated on every three days up to a final dose of one table,t three times a day at mealtimes by day 7. They will then be evaluated after two weeks and three weeks on this dose.

There are 7 visits for the study. Consent will be reviewed and signed at the beginning of visit one. All study visits include vital sign assessment, neurological exam, suicidality, tremor rating scales and Kinesia recoding. Quality of life questionnaire will be completed weekly after start. Visit one will also include collecting information on medical history, medication history and current medication. A physical exam will be done on visit one and at the end of the study. For qualifying patients, study medication will be dispensed at the end of visit one and instructions provided for titrating. Medication will be collected and counted at each visit, each arm will last for 3 weeks, with subject ET symptom assessment at week 2 and 3. After completion of week 3 assessments, all study medication will be returned, and they will change dosing to the next assigned arm where the same assessment cycle is undergone. Study medication and directions will be provided with directives to start dosing after one week wash out. After trial arm 3, subject trial participation is completed. Adverse events are assessed weekly from starting trial medication at visit one until one week after end of trial.

ELIGIBILITY:
Inclusion Criteria:

1. bilateral, largely symmetric postural or kinetic tremor involving hands and forearms that is visible and persistent. Subjects need to meet a FTMRS. Part A motor score of at least 2 ("Moderate amplitude, 0.5-1 cm, may be intermittent") in the dominant upper limb for action or postural tremor (or both).
2. additional tremor (head, voice, or lower extremity) may also be present but in the absence of abnormal posturing so as to suggest the diagnosis of dystonia.

Exclusion Criteria:

1. other abnormal neurologic signs
2. the presence of known causes of enhanced physiologic tremor, including current or recent exposure to drugs known to cause or exacerbate tremor, or the presence of a drug -withdrawal state
3. historical or clinical evidence of psychogenic tremor
4. convincing evidence of sudden onset or other evidence of stepwise deterioration
5. primary orthostatic tremor
6. isolated position-specific or task-specific tremors, including occupational tremors and primary writing tremor
7. tremor possibly or probably due to other neurological disorders (such as Parkinson's disease, cerebellar degeneration, and hyperthyroidism)
8. prior brain surgery (including deep brain stimulation of Gamma Knife treatment) for thalamotomy
9. known allergy to the study medications
10. clinically significant liver, kidney, or cardiac abnormalities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Estimated); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Fahn-Talosa-Marin rating scale (FTMRS) Part A | 11 weeks
  Comparison of placebo to each of the two medications for the sum of upper extremity postural and action tremor scores from the Fahn-Talosa-Marin rating scale (FTMRS).
  The Fahn-Tolosa-Marin Clinical Rating Scale for Tremor (FTM) has been used for essential tremor (ET), but its anchors for ratings from 0 to 4 of upper limb tremor are probably too low for patients with severe tremor (tremor amplitude >4 cm; grade 4).

CONTACTS AND LOCATIONS:
Overall Officials: Peter LeWitt, M.D., Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan, United States